CLINICAL TRIAL: NCT01514747
Title: A MRI Study of Visual and Motor Pathways in Premature Infants
Status: Completed | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: ISMRM_OU; ISMRM_2011 (Other Grant/Funding Number: ISMRM Seed Grant)
Record Dates: First submitted 2012-01-18; First posted 2012-01-23 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Premature Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ELBW infants

SUMMARY:
Approximately 30,000 babies annually are born with extremely low birth weight (ELBW) in the US. These babies often have motor and/or visual problems when they grow up. It is very important to identify high risk ELBW infants as early as possible, so that the investigators can treat them earlier to prevent poor development. Neurological examination at early age is not good enough to identify high risk ELBW infants. One the other hand, some magnetic resonance imaging (MRI) methods such as diffusion tensor imaging (DTI) and resting state functional MRI (rfMRI) have shown great sensitivity to brain injury which may cause motor and visual problems. Therefore, the investigators propose to use DTI and rfMRI on ELBW infants at a very early age to predict long-term outcome and to identify infants who are at high risk of having motor and/or visual problems when they grow up.

ELIGIBILITY:
Inclusion Criteria:

* ELBW infants with birth weight 401-1000 g (gestational age <30 weeks)

Exclusion Criteria:

* Complex congenital anomalies
* Central nervous system malformations,
* Chromosomal abnormalities, or hydrops fetalis

Ages: 2 Months to 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: ELBW infants with birth weight 401-1000 g (gestational age <30 weeks)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2011-10; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
MRI | 0

CONTACTS AND LOCATIONS:
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States